CLINICAL TRIAL: NCT02053038
Title: Prospective, Multi-center, Double Blind, Randomised Study to Test the Safety of Deferral of Stenting in Physiological Non-significant Lesions in a Clinical Population of Intermediate Stenoses Using iFR and FFR
Brief Title: Functional Lesion Assessment of Intermediate Stenosis to Guide Revascularisation
Acronym: DEFINE-FLAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 13SM1797
Record Dates: First submitted 2013-11-26; First posted 2014-02-03 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- iFR (Experimental): Treatment guided by iFR
  Interventions: Device: iFR
- FFR (Active Comparator): Treatment guided by FFR
  Interventions: Device: FFR

INTERVENTIONS:
Device: iFR — Treatment guided by instantaneous wave-free ratio
  Arms: iFR
Device: FFR — Treatment guided by Fractional Flow Reserve
  Arms: FFR

SUMMARY:
Narrowing of coronary arteries interferes with blood flow and can cause chest pain. But patients may have more than one narrowing and studies have shown that not all narrowings need to be treated. To identify the narrowings that need treating cardiologists sometimes quantify the extent of the narrowing by measuring fractional flow reserve (FFR, the ratio of the pressure in the aorta to the pressure downstream of the narrowing).This technique requires the administration of drugs that add cost and time to the procedure and in some countries are simply unavailable. As a result despite the clear health and healthcare costs benefits of FFR its use is limited to less than 5% of procedure. We have developed a new technique called the instantaneous wave-free ratio (iFR) that does not require the administration of drugs for its accurate assessment. It has been approved for use in this indication. This study aims to compare clinical outcomes of patients whose treatment has been guided by iFR to those whose treatment has been guided by FFR. If iFR is found to provide the same clinical outcomes as FFR its adoption will permit the clear benefits of this approach of identifying the coronary narrowings that really need treatment to be applicable to a much larger patient population and further improve healthcare costs.

DETAILED DESCRIPTION:
Design:

Patients with one or more coronary stenoses, in which the physiological severity from coronary angiography is in question, will be randomised 1:1 to use of the instantaneous wave free ratio (iFR) or fractional flow reserve (FFR) to guide the treatment strategy for percutaneous coronary intervention (PCI).

Aims:

To assess whether the iFR is non-inferior to FFR when used to guide treatment of coronary stenosis with PCI.

Outcome measures:

The primary endpoint will be major adverse cardiac event rate in the iFR and FFR groups at 30 days, 1, 2, and 5 years.

Population:

This will be an international multi-centre study of 2500 patients. From population estimates, 35% of the total study population will present with stable angina and 65% will have acute coronary syndrome.

Eligibility:

Patients will be eligible when the physiological severity of a stenosis within a vessel is in question. In the cases of stable angina this will be confined to the target vessel, or with acute coronary syndrome assessment this will be made in the non-culprit vessel.

Duration:

Anticipated recruitment is 12 months. Follow-up will be performed at 30 days, 1, 2 and 5 years.

Results:

Primary outcome results will be reported in Spring 2017.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age
2. Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
3. Eligible for coronary angiography and/or percutaneous coronary intervention
4. Coronary artery disease with at least 1 or more native major epicardial vessels or their branches by coronary angiogram with visually assessed de novo coronary stenosis in which the physiological severity of the lesion is in question (typically 40-70% diameter stenosis).
5. Stable angina or acute coronary syndrome (non-culprit vessels only and outside of primary intervention during acute STEMI)

Exclusion criteria:

1. Previous Coronary Artery Bypass surgery with patent grafts to the interrogated vessel
2. Significant left main stenosis (>50% narrowing)
3. Tandem stenoses separated by more than 10 mm that require separate pressure guide wire interrogation or percutaneous coronary intervention (PCI) (not to be interrogated or treated as a single stenosis)
4. Total coronary occlusions (CTOs). NOTE: Patients with CTOs can be included if i) treatment of the CTO is completed first, ii) the CTO PCI is successful, iii) the CTO PCI is successful and iii) the physiological lesion is in another vessel
5. Restenotic lesions
6. Hemodynamic instability at the time of intervention (heart rate<50 beats per minute, systolic blood pressure <90mmHg), balloon pump
7. Significant contraindication to adenosine administration (e.g. heart block, severe asthma)
8. Contraindications to PCI (percutaneous coronary intervention) or drug-eluting stent (DES) implantation
9. Heavily calcified or tortuous vessels
10. Significant hepatic or lung disease (chronic pulmonary obstructive disease), and/or malignant disease with unfavourable prognosis that may influence survival within the next 5 years
11. Pregnancy
12. STEMI (ST elevation myocardial infarction) within 48 hours of procedure
13. Severe valvular heart disease
14. ACS patients in whom more than one target vessel is present

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2021-01-19 (Estimated); Study Completion 2021-01-19 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 30 days, 1, 2 and 5 years
  Composite of death, myocardial infarction, unplanned revascularisation

SECONDARY OUTCOMES:
Death (all cause) | 30 days, 1, 2 and 5 years
Death (cardiovascular) | 30 days, 1, 2 and 5 years
Myocardial Infarction | 30 days, 1, 2 and 5 years
Repeat revascularisation | 30 days, 1, 2 and 5 years
Cost associated to iFR or FFR measurement | 30 days, 1, 2 and 5 years
  Cost associated to iFR or FFR
Quality of life assessed by EQ-5D-5L and Seattle Angina Questionnaire | 30 days, 1, 2 and 5 years
Cost savings of removing secondary investigations | 30 days, 1, 2 and 5 years
  7) Cost savings of removing secondary investigations, by assessing/treating non-culprit acute coronary syndrome (ACS) at the time of index presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Justin ER Davies, MD, Principal Investigator — Imperial College London; Javier Escaned, MD, Principal Investigator — Clinico San Carlos; Patrick Serruys, MD, Study Chair — Imperial College London; Manesh Patel, MD, Study Chair — Duke University; Sayan Sen, MD, Study Director — Imperial College London
Locations (50):
- United States (6):
  - Arnold Seto, Long Beach, California
  - John Altman, Lakewood, Colorado
  - Habib Samady, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Allen Jeremias, Stony Brook, New York
  - Manesh Patel, Durham, North Carolina
- Australia (4):
  - Sam Lehman, Adelaide
  - Darren Walters, Brisbane
  - James Sapontis, Melbourne
  - Ravinay Bhindi, Sydney
- Belgium (2):
  - Christian Vrints, Antwerp
  - Luc Janssens, Bonheiden
- Ahmed Khashaba, Cairo, Egypt
- Mika Laine, Helsinki, Finland
- Germany (4):
  - Florian Krackhardt, Berlin
  - Olaf Going, Berlin
  - Waldemar Bojara, Koblenz
  - Tobias Haerle, Oldenburg
- Italy (3):
  - Ciro Indolfi, Catanzaro
  - Giampaolo Nicolli, Rome
  - Flavio Ribichini, Verona
- Japan (5):
  - Hiroaki Takashima, Aichi
  - Hiroyoshi Yokoi, Fukuoka
  - Yuetsu Kikuta, Fukuyama
  - Hitosh Matsuo, Gifu
  - Nob Tanaka, Tokyo
- Andrejs Erglis, Riga, Latvia
- Netherlands (3):
  - Jan Piek, Amsterdam
  - Niels Van Royen, Amsterdam
  - Martijn Meuwissen, Breda
- Portugal (3):
  - Hugo Vinhas, Almada
  - Sergio Baptista, Amadora
  - Pedro Canas Silva, Lisbon
- Ali Alghamadi, Riyadh, Saudi Arabia
- Farrel Hellig, Johannesburg, South Africa
- South Korea (4):
  - Chang-Wook Nam, Daegu
  - Joon-Hyung Doh, Daehwa
  - Bon-Kwon Koo, Seoul
  - Eun-Seok Shin, Ulsan
- Spain (3):
  - Salvatore Brugaletta, Barcelona
  - Clinico San Carlos, Madrid
  - Eduardo Alegria, Madrid
- Murat Sezer, Istanbul, Turkey (Türkiye)
- United Kingdom (7):
  - Kare Tang, Basildon
  - Suneel Talwar, Bournemouth
  - Andrew Sharp, Exeter
  - Imperial College London, London
  - Ranil De Silva, London
  - Rajesh Kharbanda, Oxford
  - Robert Gerber, St Leonards

REFERENCES:
- [Derived] Escaned J, Travieso A, Dehbi HM, Nijjer SS, Sen S, Petraco R, Patel M, Serruys PW, Davies J; DEFINE FLAIR Investigators. Coronary Revascularization Guided With Fractional Flow Reserve or Instantaneous Wave-Free Ratio: A 5-Year Follow-Up of the DEFINE FLAIR Randomized Clinical Trial. JAMA Cardiol. 2025 Jan 1;10(1):25-31. doi: 10.1001/jamacardio.2024.3314. PMID 39412778
- [Derived] Eftekhari A, Holck EN, Westra J, Olsen NT, Bruun NH, Jensen LO, Engstrom T, Christiansen EH. Instantaneous wave free ratio vs. fractional flow reserve and 5-year mortality: iFR SWEDEHEART and DEFINE FLAIR. Eur Heart J. 2023 Nov 1;44(41):4376-4384. doi: 10.1093/eurheartj/ehad582. PMID 37634144
- [Derived] Kim CH, Koo BK, Dehbi HM, Lee JM, Doh JH, Nam CW, Shin ES, Cook CM, Al-Lamee R, Petraco R, Sen S, Malik IS, Nijjer SS, Mejia-Renteria H, Alegria-Barrero E, Alghamdi A, Altman J, Baptista SB, Bhindi R, Bojara W, Brugaletta S, Silva PC, Di Mario C, Erglis A, Gerber RT, Going O, Harle T, Hellig F, Indolfi C, Janssens L, Jeremias A, Kharbanda RK, Khashaba A, Kikuta Y, Krackhardt F, Laine M, Lehman SJ, Matsuo H, Meuwissen M, Niccoli G, Piek JJ, Ribichini F, Samady H, Sapontis J, Seto AH, Sezer M, Sharp ASP, Singh J, Takashima H, Talwar S, Tanaka N, Tang K, Van Belle E, van Royen N, Vinhas H, Vrints CJ, Walters D, Yokoi H, Samuels B, Buller C, Patel MR, Serruys PW, Escaned J, Davies JE. Sex Differences in Instantaneous Wave-Free Ratio or Fractional Flow Reserve-Guided Revascularization Strategy. JACC Cardiovasc Interv. 2019 Oct 28;12(20):2035-2046. doi: 10.1016/j.jcin.2019.06.035. PMID 31648764
- [Derived] DEFINE-FLAIR Trial Investigators; Lee JM, Choi KH, Koo BK, Dehbi HM, Doh JH, Nam CW, Shin ES, Cook CM, Al-Lamee R, Petraco R, Sen S, Malik IS, Nijjer SS, Mejia-Renteria H, Alegria-Barrero E, Alghamdi A, Altman J, Baptista SB, Bhindi R, Bojara W, Brugaletta S, Silva PC, Di Mario C, Erglis A, Gerber RT, Going O, Harle T, Hellig F, Indolfi C, Janssens L, Jeremias A, Kharbanda RK, Khashaba A, Kikuta Y, Krackhardt F, Laine M, Lehman SJ, Matsuo H, Meuwissen M, Niccoli G, Piek JJ, Ribichini F, Samady H, Sapontis J, Seto AH, Sezer M, Sharp ASP, Singh J, Takashima H, Talwar S, Tanaka N, Tang K, Van Belle E, van Royen N, Vinhas H, Vrints CJ, Walters D, Yokoi H, Samuels B, Buller C, Patel MR, Serruys P, Escaned J, Davies JE. Comparison of Major Adverse Cardiac Events Between Instantaneous Wave-Free Ratio and Fractional Flow Reserve-Guided Strategy in Patients With or Without Type 2 Diabetes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2019 Sep 1;4(9):857-864. doi: 10.1001/jamacardio.2019.2298. PMID 31314045
- [Derived] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458